CLINICAL TRIAL: NCT04244500
Title: Burden of Influenza at Emergency Department (ED) Level in European Countries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Collaborators: Klinikum Ernst von Bergmann Potsdam (Unknown); Klinikum Suedstadt, Rostock (Unknown); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Dr. med. Micha Loebermann, Deputy head of Department, University of Rostock
Other Study IDs: UMR893958
Record Dates: First submitted 2020-01-12; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Influenza, Human
Keywords: emergency room; epidemiology
MeSH Terms: conditions — Influenza, Human; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Influenza: Influenza testing
  Interventions: Procedure: swab sampling

INTERVENTIONS:
Procedure: swab sampling — Multiplex polymerase chain reaction assay for organisms of upper respiratory tract infections

SUMMARY:
This study plans to conduct enhanced influenza surveillance at a hospital emergency department level independent of underlying influenza-like symptoms.

DETAILED DESCRIPTION:
Study objectives

Primary:

- Measure the proportion of non-traumatic emergency department (ED) visits infected with influenza during the peak of the influenza season

Secondary:

* Describe the demographic and medical profile of influenza-related and non-influenza-related visits
* Identify socio-demographic or other risk factors associated with ED visit outcome
* Describe the influenza positivity rate among ED visits for different causes
* Measure the proportion of influenza positive patients without classical ILI symptoms

ELIGIBILITY:
Inclusion Criteria:

* All adult patients seeking care at participating ED during the influenza season
* Participants and/or guardian providing informed consent and/or assent, as appropriate, to participate.

Exclusion Criteria:

* Individuals reporting having suffered a traumatic injury without other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients seeking care at the emergency department of participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
influenza status at admission to ED (positive vs. negative) | at admission to ED
  proportion of non-traumatic emergency department (ED) visits infected with influenza during the peak of the influenza season

SECONDARY OUTCOMES:
demographic and medical profile | at admission to ED
  demographic and medical profile of influenza-related and non-influenza-related visits
socio-demographic or other risk factors | at admission to ED
  Identify socio-demographic or other risk factors associated with ED visit outcome
influenza without classical symptoms of influenza-like illness | at admission to ED
  Measure the proportion of influenza positive patients without classical ILI symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rostock, Rostock, Germany

IPD SHARING:
Plan to Share IPD: Undecided